CLINICAL TRIAL: NCT01800552
Title: Ultrasound Detection of Peripheral IV Infiltration
Status: Completed | Type: Observational
Sponsor: ivWatch, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: IVWUS-001
Record Dates: First submitted 2013-02-22; First posted 2013-02-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Infiltration; IV Infiltration
Keywords: Infiltration; Extravasation; Leaking; PIV Infiltration; IV Infiltration; Ultrasound Detection of Infiltration; Ultrasound Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Intentional infiltration of a peripheral IV site — An intentional infiltration of isotonic saline solution is performed by pushing the needle through the vein wall into the subcutaneous tissue. A total volume less than or equal to 5 cc of saline is infiltrated into the tissue.

SUMMARY:
The purpose of this study is to determine whether commercial ultrasound imaging systems can discern normal from infiltrated tissue near a peripheral intravenous site.

DETAILED DESCRIPTION:
Peripheral intravenous (PIV) therapy is one of the most common invasive procedures performed in US hospitals. A majority of hospital patients require intravenous therapy each year in the United States. Despite widespread use, a number of potential complications can occur during PIV therapy. One of the most common causes of IV complications is IV infiltration or extravasation. Infiltration is the leakage of non-vesicant fluids like saline into the surrounding tissue. Extravasation is the leakage of vesicant fluids, which include cytotoxic drugs, intravenous nutrition, and calcium, potassium, and bicarbonate solutions. If not detected and corrected early, infiltration and extravasation can lead to significant complications such as severe inflammation, compartment syndrome, and skin necrosis.

ivWatch, LLC has developed an investigational device that may detect IV infiltration and extravasation occurrences using a near infrared light sensor. Previous studies have evaluated the performance of the ivWatch device by comparing to a nurse's diagnosis. The nursing standard of care relies on tactile and visual indicators to diagnose an infiltration event. The ivWatch product often signals an infiltration event before these indicators are apparent to clinicians. Consequently, comparisons to the nurse's diagnosis often lead to questionable false positives for the ivWatch device. A better reference is required to evaluate the performance of the ivWatch device.

The purpose of this research study is to evaluate the ability of ultrasound to detect PIV infiltrations. Ultrasound is a depth-resolved imaging technique for evaluating tissue microstructure. Researchers have used ultrasound to examine exogenous fluids injected into cutaneous and subcutaneous tissue. Ultrasound has been used to detect small volumes of fluids such as cosmetic fillers and subcutaneous injections. These studies suggest ultrasound may be a potential reference standard for future evaluation of ivWatch devices.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* signed consent
* health form approved by professional practitioner

Exclusion Criteria:

* abnormal bleeding or hemophilia
* absence of sensation in arms
* anemia
* cardiopulmonary disorders
* clotting disorders
* dehydration
* dizziness or fainting
* hepatitis
* high blood pressure (>160 systolic or > 115 diastolic)
* HIV / AIDS
* immune deficiency disorders
* known history of difficult venous access
* lymphedema
* major surgery or scar tissue which would complicate venous access
* recent radiation or chemotherapy
* received IV therapy in past 30 days
* history of seizures
* history of strokes
* sick or had infection in past 30 days
* high temperature (>99.6F)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers (18 years or older) that were friends, family members, or employees of ivWatch, LLC participated in this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Test diagnostic performance of ultrasound imaging for detection of peripheral IV infiltration. | Within 15 minutes of intentional PIV infiltration
  Ultrasound images are acquired before and after the induced infiltration on the test arm. Two additional ultrasound images are acquired from the normal control arm. At the end of the study, the before and after images from the test and control arms are evaluated and classified by clinicians blinded to the state of the tissue. Sensitivity and specificity metrics are used to evaluate the performance of ultrasound imaging for assessing peripheral IV infiltration.

CONTACTS AND LOCATIONS:
Overall Officials: Garret T Bonnema, Ph.D., Principal Investigator — ivWatch, LLC
Locations (1):
- ivWatch,LLC, Williamsburg, Virginia, United States